CLINICAL TRIAL: NCT07021560
Title: A Double Masked, Randomised, Longitudinal Comparative Study to Evaluate the Wearability and Myopia Progression of ZEISS MyoCare Spectacle Lenses Versus Two ZEISS Single Vision Spectacle Lenses in Children With Myopia
Brief Title: Wearability of and Myopia Progression With ZEISS MyoCare Spectacle Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZEISS Vision Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28/CV-MHN2
Record Dates: First submitted 2025-05-16; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Myopia
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SV 1 (Active Comparator): Single vision lenses
  Interventions: Device: ZEISS SV RX SPH 1.5
- SV 2 (Active Comparator): Single vision lenses
  Interventions: Device: ZEISS Clearview
- MyoCare (Experimental): ZEISS MyoCare spectacle lenses
  Interventions: Device: ZEISS MyoCare spectacle lenses

INTERVENTIONS:
Device: ZEISS MyoCare spectacle lenses — Spectacle lenses with conventional power profile including myopia control design.
  Arms: MyoCare
Device: ZEISS SV RX SPH 1.5 — Commercially available single vision
  Arms: SV 1
Device: ZEISS Clearview — Commercially available single vision
  Arms: SV 2

SUMMARY:
This is a clinical trial evaluating the wearability and effectiveness of three types of ZEISS spectacle lenses in controlling myopia progression. This study compares ZEISS MyoCare spectacle lenses with two types of single-vision spectacle lenses over a 6-month period. This trial aims to evaluate how well these lenses are worn and their impact on myopia progression, including changes in axial length and refractive error.

Participants will be randomly assigned to wear one of three types of ZEISS spectacle lenses. The study will require five visits to the eye clinic over a 6-month period and two virtual follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* be accompanied by a parent or guardian who is able to read and comprehend Vietnamese/English and sign a record of informed consent/assent;
* at baseline, be within the age range of 7 to 13 years old inclusive;
* be diagnosed as myopic having cycloplegic spherical equivalent between -0.75 dioptre (D) and -5.00 dioptre (D);
* astigmatism ≤1.50D;
* anisometropia of not more than 1.50D;
* be willing to comply with the wearing of clinical trial spectacles and clinical trial visit schedule as directed by the investigator;
* have ocular findings deemed to be normal;
* vision correctable to at least 0.8 or better in each eye with spectacles.

Exclusion Criteria:

* Any pre-existing systemic or ocular condition, including infection or disease that is likely to affect visual acuity and refractive error;
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology in an adverse or beneficial manner at enrolment and/or during the clinical trial. NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.
* History of eye trauma or eye surgery
* Amblyopia
* Anisometropia of not more than 1.50D
* Strabismus
* History of use of myopia control interventions such as Orthokeratology or atropine 3 months prior to commencement of this trial.
* Known allergy or intolerance to ingredients to cycloplegic eye-drops.
* Currently enrolled in another clinical trial.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Wearability | Day 1 At dispensing visit, 3 months and 6 months visits
  Visual acuity with study spectacle lenses
Wearability | Day 1 At dispensing visit, 1-week and 2-week visits, and 3 months and 6 months visits
  Subjective responses measured by a wearability questionnaire (scale 1-10, with 1 being the worst and 10 being the best) regarding study spectacle lenses wear
Wearability | At 1-week, 2-week, 3 months and 6 months visits
  Compliance (lens wearing time, hr/day) to study spectacle lenses wear

SECONDARY OUTCOMES:
Myopia progression | At baseline and 6 months visits
  The 6 monthly myopia progression measured by change in spherical equivalent from baseline for each of the study groups.
Myopia progression | At baseline, 3 months, and 6 months visits
  The 6 monthly myopia progression measured by change in axial length from baseline for each of the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hoang Viet Vu, MD, Principal Investigator — Hanoi Eye Hospital 2
Locations (1):
- Hanoi Eye Hospital 2, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No